CLINICAL TRIAL: NCT07065968
Title: Teriflunomide and High-dose Dexamethasone vs High-dose Dexamethasone Alone as First-line Treatment for Newly Diagnosed Adult Primary Immune Thrombocytopenia: A Prospective, Multicenter, Randomized Trial
Brief Title: The Efficacy and Safety of Combined Teriflunomide and High-dose Dexamethasone in Newly Diagnosed Primary Immune Thrombocytopenia (TEMPO-2)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University Health Science Center (Other); Cisen Pharmaceutical CO., LTD. (Industry)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TY2025006
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — teriflunomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teriflunomide plus Dexamethasone (Experimental): Oral Teriflunomide was given at a dose of 14 mg once daily for 24 weeks, and dexamethasone was given at a dose of 40mg orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4). Nonresponsive participants with platelets less than 30 x10^9/L or with active bleeding were allowed to repeat the 4-day course of dexamethasone treatment.
  Interventions: Drug: Teriflunomide; Drug: Dexamethasone
- Dexamethasone (Active Comparator): Dexamethasone was given at a dose of 40mg, orally once per day for 4 consecutive days (Days 1, 2, 3, and 4). Nonresponsive participants with platelets less than 30 x10^9/L or with active bleeding were allowed to repeat the 4-day course of dexamethasone treatment.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Teriflunomide — Teriflunomide 14 mg orally once daily for 24 weeks.
  Arms: Teriflunomide plus Dexamethasone
Drug: Dexamethasone — Dexamethasone 40 mg orally once daily for four consecutive days.

SUMMARY:
A multicenter, open-label, randomized study to report the efficacy and safety of teriflunomide plus high-dose dexamethasone compared to high-dose dexamethasone monotherapy for the first-line treatment of adults with newly diagnosed primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators are undertaking a parallel-group, multicenter, randomized controlled trial of 132 adults with ITP in China. Patients were randomized to teriflunomide plus high-dose dexamethasone and high-dose dexamethasone monotherapy group. Platelet count, bleeding, and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years;
2. Newly diagnosed, treatment naïve ITP patients;
3. Patients with a platelet count <30 x10^9/L or a platelet count <50 x10^9/L with bleeding manifestations at the enrollment;
4. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Secondary ITP such as drug-related thrombocytopenia, viral infection (HIV, hepatitis B virus, or hepatitis C virus);
2. Pre-existing acute or chronic liver disease, or ALT/AST greater than 2 times the upper limit of normal (ULN);
3. Severe cardiac, renal, hepatic, or respiratory insufficiency;
4. Severe immunodeficiency;
5. Pregnancy or lactation;
6. Active or a history of malignancy;
7. Active infection requiring systemic therapy;
8. Myelodysplastic syndrome, aplastic anemia, or myelofibrosis;
9. A known diagnosis of other autoimmune diseases;
10. Patients who are deemed unsuitable for the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2027-09-10 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Sustained response | Week 24
  Sustained response was defined as a platelet count ≥ 30 x10^9/L and at least a 2-fold increase of the baseline count in the absence of bleeding and rescue therapy for at least three of the four visits of the last 8 weeks of treatment.

SECONDARY OUTCOMES:
Initial response | Week 4
  The number of participants with achievement of CR or R at 4 weeks. Complete response (CR) was defined as a platelet count ≥ 100 x10^9/L and absence of bleeding. Response (R) was defined as a platelet count ≥ 30 x10^9/L and at least a 2-fold increase of the baseline count and absence of bleeding. No response was defined as a platelet count of less than 30 x10^9/L, or less than two times increase from baseline platelet count, or bleeding.
Time to response | Week 24
  The time from treatment initiation to time of achievement of CR or R.
Duration of response | Week 24
  The time from the achievement of a CR or R to the loss of CR or R.
Bleeding events | Week 24
  Clinically significant bleeding was assessed using the World Health Organization (WHO) bleeding scale.
Adverse events | Week 24
  Adverse events (AEs) were reported and graded according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
Health-related quality of life (HRQoL) | Week 24
  ITP-patient assessment questionnaire (ITP-PAQ) was used to assess the HRQoL before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Hui Zhang, MD, Principal Investigator — Peking University Institute of Hematology, Peking University People's Hospital
Locations (3):
- China (3):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No